CLINICAL TRIAL: NCT03432715
Title: Approaches to Enhancing Wellness Policy Implementation in Schools to Promote Healthy Behaviors and Prevent Obesity
Brief Title: Wellness Champions for Change
Acronym: WCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); University of Maryland, College Park (Other); Boise State University (Other); University of Southern California (Other); Cornell University (Other)
Responsible Party: Principal Investigator, Erin Hager, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: HP-00067626
Record Dates: First submitted 2018-02-02; First posted 2018-02-14 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Obesity, Childhood
Keywords: School; Policy; Nutrition; Physical Activity; Local Wellness Policy
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: A portion of participating schools will receive a Student Wellness Champion curriculum, training for their wellness team, as well as technical assistance provided by a Wellness Specialist (WCC-S Group). Other participating schools will only receive the training and technical assistance (WCC Group) and some will solely receive resources (Control Group). The process to determine which school receives which intervention is completely random, and will not be decided until after baseline data collection.
Who Masked: Outcomes Assessor
Masking Description: All data collectors are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wellness Champions for Change + Students (Experimental): Schools randomized to the WCC+S arm will receive both the Teacher Intervention and the Student Wellness Champion Intervention.
  Interventions: Behavioral: Student Wellness Champions; Behavioral: Teacher Wellness Champions
- Wellness Champions for Change (Experimental): Schools randomized to the WCC+S arm will receive only the Teacher Intervention.
  Interventions: Behavioral: Teacher Wellness Champions
- Control (No Intervention): The control group will not receive either intervention. Schools will be given a modified SWC curriculum as well as the teacher training at the end of the data collection period.

INTERVENTIONS:
Behavioral: Student Wellness Champions — Student Wellness Champions participate in a training to, develop a rapport, and build trust with the wellness specialist. SWCs will meet once/week during lunch. The SWC's will receive a health education/ health literacy curriculum in order to be well-versed on the importance of being active and eating healthy foods and how to communicate health information to key stakeholders to enact policy change and to fellow students to enact behavior change. These students will work with the Wellness Specialist and Wellness Champion to implement wellness policies and practices.
  Target policies/practices will be presented as a menu of options. The mechanisms used to enact change are based in the tenets of health literacy anchored in nutrition and PA promotion. Components of the curriculum include raising awareness of school system's local wellness policies and improving student skills surrounding the five standards of health literacy, using examples/activities linked to the local wellness policy.
  Arms: Wellness Champions for Change + Students
Behavioral: Teacher Wellness Champions — Schools will be asked to identify a Wellness Champion (WC), someone at the school who is passionate about creating a healthy school environment. All WC's will be asked to attend a Wellness Champions for Change (WCC) training, led by a Wellness Specialist (health educator part of our study team). The WC's will learn about the skills necessary to make health promoting changes to the School Environment.
  Following the WCC training, the Wellness Champion will receive technical assistance from the Wellness Specialist. The Wellness Specialist will work with the Wellness Champion and the school's Wellness Team to conduct a needs assessment, and develop and implement a school action plan. The Wellness Specialist will provide support and resources to the Wellness Champion and the school to help them work towards their goals. All Wellness Champions in a given school system will meet monthly, as a group, with their Wellness Specialist to discuss progress, pitfalls, and successes.
  Arms: Wellness Champions for Change; Wellness Champions for Change + Students

SUMMARY:
The Wellness Champions for Change (WCC) study aims to reduce pediatric obesity among students who attend schools in Maryland by training teacher and student-led wellness teams to increase opportunities for physical activity and healthy eating at school.

The study uses a cluster randomized design to allocate 6 schools (3 elementary, 3 middle) in 5 school systems to one of 3 arms: "A" (teacher and student training), "B" (teacher training only), and "C") (delayed teacher training/control). Approximately 36 3rd/6th graders and their caregivers ("evaluation cohort"), 15 4th/7th graders ("student leaders"), and 20 teachers from each school will be recruited in the spring before the intervention. All schools will identify a teacher "Wellness Champion" who will coordinate intervention activities. In "A" and "B" schools, wellness champions will attend a training to learn how to build a wellness team and create more opportunities for students to make healthy choices. In "A" schools, student leaders ("Student Wellness Champions") will meet weekly during lunch with a health educator to receive training as peer leaders and help the Wellness Champion with wellness initiatives. Student leaders in "B" and "C" schools will receive a monthly general Adolescent Health Curriculum. To assess the impact of the teacher and student-led interventions, the evaluation cohort will be followed for 2.5 years, with measures including: anthropometry (height/weight), 7-day accelerometry (physical activity), and validated questionnaires to assess healthy eating. Student leaders will be followed for 1.5 years to assess the impact of their participation, with measures including: anthropometry, 7-day accelerometry, validated questionnaires to assess healthy eating, and validated questionnaires and focus groups to assess leadership/advocacy skills. Teachers will complete validated questionnaires to investigate their perceptions of the school environment, classroom practices, and role modeling skills. Prior to data collection and analysis, participants will be assigned an identification number, and all documents linking participant information to identification numbers will be locked/ password-protected.

DETAILED DESCRIPTION:
The long-term goal of this project is to create health promoting school environments that support healthy growth and development of children in order to prevent obesity. The approach for creating health promoting school environments involves the school-level implementation of existing Local Wellness Policies (LWPs). Implementation science suggests that policy implementation may occur through diffusion ("letting it happen"), dissemination ("helping it happen"), or implementation ("making it happen"). Since LWPs were initially mandated in 2006, most school systems have relied on a diffusion or dissemination approach to LWP implementation, leading to limited implementation on the school-level. We propose a school-level LWP implementation strategy ("making it happen") that relies on educating/training teachers and students to be wellness champions. Through this proposed study, the impact of a school-level intervention to enhance LWP implementation (WCC) and the added benefit of training students to be wellness champions (WCC-students, "WCC-S") on student-level outcomes [diet, physical activity (PA), and obesity] will be examined through a randomized controlled trial.

Objectives are presented at the student and student wellness champion level:

Student Objectives:

Aim 1: To determine the impact of a school-based intervention ("Wellness Champions for Change" (WCC)) to enhance implementation of LWPs, on health behaviors (diet and PA) and weight status of elementary and middle school students through a randomized controlled trial.

Hypothesis 1: WCC will have a positive impact on health behaviors of students, compared to control.

Aim 2: To examine the added impact of a student-led school-based intervention ("Wellness Champions for Change-Students" (WCC-S) on health behaviors (diet and PA) and weight status of elementary and middle school students through a randomized controlled trial.

Hypothesis 2: WCC+WCC-S will have a greater impact on health behaviors of students, compared to WCC and control.

Aim 3: To examine factors in the home and school-neighborhood environments that moderate the impact of WCC/WCC-S on health behavior (diet and PA) and weight status change of elementary/middle school students.

Hypothesis 3: Students living in a moderately health-promoting home and school-neighborhood environment will experience a greater change in health behaviors when exposed to WCC or WCC+WCC-S compared to students in high or low health-promoting environments.

Aim 4: To examine the reach and fidelity of WCC and WCC-S when disseminated via eXtension through an online continuing education credit model for teachers and a toolkit for students.

Hypothesis 4: WCC and WCC-S dissemination schools will experience positive changes in LWP implementation.

Student Wellness Champion Objectives:

One part of our study involves developing a Student Wellness Champions curriculum (WCC-S group) to train 5th and 8th graders in diverse schools across Maryland to make policy and environmental changes that create a "health-promoting environment" in their schools. We plan to evaluate individual and organizational outcomes for the 5th and 8th grade student wellness champions:

Aim 1: To assess the individual effectiveness of WCC-S to improve student wellness champions youth advocacy, health literacy and public health literacy constructs, and changes in diet and physical activity behaviors and/or weight status compared to control students.

Aim 2: To asses organizational effectiveness of WCC-S to improve school level LWP implementation and environmental change compared to control or WCC-only schools.

Aim 3: To describe reach, adoption, implementation, and maintenance factors including- reach and representativeness of student champions, extent to which the intervention reaches other students in WCC-S schools, representativeness of adopting schools compared to non-adopting schools, implementation fidelity, barriers and challenges of implementation of training and goal achievement, which intervention aspects (if any) are institutionalized.

A portion of participating schools will receive a Student Wellness Champion curriculum, training for their wellness team, as well as technical assistance provided by a Wellness Specialist (WCC-S Group). Other participating schools will only receive the training and technical assistance (WCC Group) and some will solely receive resources (Control Group). The process to determine which school receives which intervention is completely random, and will not be decided until after baseline data collection.

In the spring prior to the intervention, all participating schools will be asked to select a group of about 15 students (4th graders in elementary schools, 7th graders in middle schools) to be a part of a Health Leader group that begins the following year (when the same students are 5th graders in elementary, 8th graders in middle school). Students can either be nominated by teachers or write a few sentences on why the student thinks it is important to make his/her school a healthier place. At the beginning of the next school year, the health leaders that attend schools randomized to WCC-S will become Student Wellness Champions. These students will meet with a Wellness Specialist (member of our project team) once a week during lunch to receive a health education/ health literacy curriculum in order to be well-versed on the importance of being active and eating healthy foods, and how to communicate health information to key stakeholders (administration and teachers) to enact policy change and to fellow students to enact behavior change. These students will work with the Wellness Specialist and staff members from their school to implement wellness policies and practices. Health leaders that attend schools randomized to the WCC or control schools will remain Health Leaders, and will have the opportunity to participate in an Adolescent Health Curriculum, taught by the Wellness Specialist, during their 5th or 8th grade year. These students will meet once a month, during lunch, and the curriculum will focus on general public health topics including dental health, stress management and hygiene. At the end of the year, participants will also have the opportunity to participate in a public health leadership workshop.

Schools randomized to WCC-S and WCC will select a teacher to become the Wellness Champion (WC). This person may be a teacher or other school leader (nurse, counselor, etc.) who is passionate about creating a healthy school environment. The wellness champions will attend a Wellness Champions for Change training prior to the start of the intervention. During the training, the Wellness Champion will work with a Wellness Specialist to set achievable LWP implementation goals and design a plan for implementing those goals over the academic year. Furthermore, this training will equip the Wellness Champion to build a school-level wellness team, assess the school's wellness environment, develop, monitor, and report a school LWP action plan, and conduct wellness activities that align with the LWP.

Following the training, the Wellness Champion will work with the school's wellness team to develop and implement a school LWP action plan. All Wellness Champions in a given school system will meet monthly, as a group, with the Wellness Specialist to discuss progress, pitfalls, and successes (bi-monthly in-person and/or bi-monthly by phone). In addition, all Wellness Champions will receive year-long technical assistance from the Wellness Specialist that focuses on implementing and monitoring LWP's at the school-level. The WCC intervention will formally last for one school year, with schools continually followed for an additional year to assess sustainability.

In order to measure the success of the intervention, evaluations on a group of 36 students from all participating schools will be conducted (recruited as 3rd grade students in elementary school and 6th grade students in middle schools). These students will become members of the Evaluation Cohort, and will be asked to be followed for 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Student attends a school that the Wellness Champions for Change Study has selected for the intervention year
* Student is enrolled in the correct grade during spring recruitment
* Student has the ability to read and write in English
* Student has the ability to complete grade level surveys independently
* Student has a participant caregiver

Exclusion Criteria:

* Student has a health problem that would interfere with participation in physical education classes
* Student is enrolled in a special education class (Health Leaders/SWC only)
* Another student in the same grade living in the same household or who shares the same primary caregiver is already enrolled in the study (Evaluation Cohort Only)

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2773 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Overweight/obesity | 5 years
  BMI-for-age z-score (calculated based on measured height and weight; self-reported gender and date of birth)
In-school diet behaviors | 5 years
  Dietary screener (Patterns of Diet at School: PODS)
Minutes per day in Moderate-Vigorous Physical Activity | 5 years
  Accelerometry (Actical); placed on the ankle

SECONDARY OUTCOMES:
School environment specific to healthy eating and physical activity | 5 years
  School audit
School environment specific to healthy eating and physical activity | 5 years
  Survey (Perceptions of the Environment At School: PEAS)

CONTACTS AND LOCATIONS:
Overall Officials: Erin R Hager, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuhn AP, Choudhary A, Zemanick A, Lane H, Armstrong B, Wang Y, Deitch R, Hager ER. Student perceptions of U.S. based school day physical activity best practices in relation to accelerometer-based sedentary behavior and activity. Prev Med Rep. 2024 Dec 16;49:102944. doi: 10.1016/j.pmedr.2024.102944. eCollection 2025 Jan. PMID 39807184
- [Derived] Pulling Kuhn A, Kim E, Lane HG, Wang Y, Deitch R, Turner L, Hager ER, Parker EA. Associations between elementary and middle school teachers' physical activity promoting practices and teacher- and school-level factors. Int J Behav Nutr Phys Act. 2021 May 19;18(1):66. doi: 10.1186/s12966-021-01129-4. PMID 34011376